CLINICAL TRIAL: NCT04315766
Title: Optimised Lung Cancer Screening to Prevent Cardiovascular and Pulmonary Diseases Coupled With Primary Prevention
Acronym: SMAC-1
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istituto Clinico Humanitas (Other)
Collaborators: Ospedale San Raffaele (Other)
Responsible Party: Sponsor
Other Study IDs: 2123
Record Dates: First submitted 2019-01-10; First posted 2020-03-20 (Actual); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Lung Cancer; Cardiovascular Disease (CVD); Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Cancer risk prevention; Cancer risk reduction; Cardiovascluar disease prevention; microRNAs; COPD prevention; Lung cancer circulating biomarkers; Lung cancer screening; Minimally invasive surgery; Low Dose Computed Tomography (LDCT)
MeSH Terms: conditions — Lung Neoplasms; Cardiovascular Diseases; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This project aims to implement a health prevention program for smokers or former smokers including early detection of lung cancer, cardiovascular disease (CVD) and chronic obstructive pulmonary disease (COPD). The clinical activity is completed by a pre-clinical evaluation of molecular bio-markers of early diagnosis of these diseases, with the aim of strengthening the sensitivity and specificity of the screening program.

The project also includes a cost-effectiveness assessment to validate the feasibility of the program.

Since lung cancer, CVD and COPD are among the deadliest smoking-related pathologies, the program includes actions aimed at raising awareness among primary care physicians, increasing the smoking cessation rate of participating subjects to improve quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 55 years old and exposure to smoking more than 30 packs-year; which corresponds to 6-year risk of lung cancer, calculated according to the plco score (≥ 2%).
* Smoker or former smoker Former smokers must have ceased smoking within the 15 years prior to enrollment in the study.
* Absence of symptoms of lung cancer such as worsening of cough, hoarseness, hemoptysis and weight loss.

Exclusion Criteria:

* Previous diagnosis of lung cancer.
* Positive extrapulmonary cancer history in the last 5 years (excluding in situ tumors or skin epidermoid tumor).
* Performing a chest CT scan in the last 18 months.
* Severe lung or extrapulmonary diseases that may preclude or invalidate appropriate therapy in case of diagnosis of malignant pulmonary neoplasia.

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population should have the following inclusion criteria:
  Inclusion Criteria:
  * Age ≥ 55 years old and exposure to smoking more than 30 packs-year; which corresponds to 6-year risk of lung cancer, calculated according to the plco score (≥ 2%).
  * Smoker or former smoker Former smokers must have ceased smoking within the 15 years prior to enrollment in the study.
  * Absence of symptoms of lung cancer such as worsening of cough, hoarseness, hemoptysis and weight loss.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2018-10-10 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
To implement the screening program combining lung cancer, CVD and COPD prevention | from 10 Oct 2018 to 10 Oct 2021
  Subjects with increased risk for lung cancer, selected through an epidemiological questionnaire, sign the informed consent and their blood is collected. They then undergo LDCT and an interview at the anti-smoking center. CTs presenting with at least one non-calcified nodule are managed according to dedicated diagnostic algorithm. Nodules indicative of lung cancer will be studied with preoperative diagnosis, with surgical resection preferably performed with a minimally invasive approach. Multimodality treatment is indicated in advanced stage of disease. Subjects with normal findings are scheduled for annuals CT scan for two additional years. Cardiovascular risk will be assessed with the use of the atherosclerotic cardiovascular disease (ASCVD) score, recommended by the American College of Cardiology/American Heart Association, integrated with Reynold risk score and CAC score. The CAC score, calculated on LDCT, is used to quantify the presence of calcium through the coronary system.

SECONDARY OUTCOMES:
Validation of circulating markers to enhance LDCT sensitivity and specificity of the screening for lung cancer, CVD and COPD early detection. | from 10 Oct 2018 to 10 Oct 2021
  Ten ml of blood is collected before LDCT, for plasma and white blood cells. For lung cancer patients, blood is collected before treatment, at 1-6-12 months after treatment, to analyse markers for minimal residual disease or early recurrence.
  We will perform:
  * CTC identification and genomic analysis. Patients are considered CTCs positive based on cytopathology of the isolated cells and detection of characteristic malignant features.
  * Evaluation of Serum of PTX3, measured with an original sandwich enzyme-linked immunosorbent assay (ELISA)
  * Circulating microRNA profiling. A custom panel of 6 specific microRNAs identified in a previous study on Karolinska cohort and correlating with increase/reduction risk of CVD Mayor adverse cardiovascular events MACE will be tested in 2000 patients.
  * IL-2, IL-8, CRP, IL-5 and Eosinophils analyses. Interleukin-2 and-8, C-reactive protein, interleukiine-5 and eosinophils concentrations in blood are measured with ELISA kits.
Cost benefit analysis of LC screening program | from 10 Oct 2018 to 10 Oct 2021
  Cost-benefit analysis of the prevention program. Direct and indirect costs associated with diagnosis and treatment of smoking-related diseases will be compared to those of a control group with disease detected after the appearance of pulmonary symptoms. The incremental cost effectiveness ratio will be evaluated in terms of QUALYS (quality of life adjusted years saved).

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Clinico Humanitas, Rozzano, Milano, Italy

IPD SHARING:
Plan to Share IPD: No